CLINICAL TRIAL: NCT00402506
Title: MEND-CABG II: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Evaluate the Cardioprotective Effects of MC-1 in Patients Undergoing High-Risk CABG Surgery
Brief Title: A Safety and Efficacy Study to Confirm the Cardioprotective Effects of MC-1 in Patients Undergoing High-Risk CABG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medicure (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06004
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2007-11-16 (Estimated); Status verified 2007-11

CONDITIONS: Coronary Artery Bypass Graft Surgery; Myocardial Ischemia; Reperfusion Injury
Keywords: coronary; surgery; ischemia; reperfusion injury; cardiac; heart; neurological; cardiopulmonary bypass; cardioprotection; myocardium; myocardial; myocardial revascularization
MeSH Terms: conditions — Myocardial Ischemia; Reperfusion Injury; Ischemia; Neurologic Manifestations | interventions — Pyridoxal Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: (MC-1) Pyridoxal 5'-phosphate

SUMMARY:
The purpose of this study is to determine the effect of MC-1 on the combined incidence of cardiovascular death and nonfatal myocardial infarction (MI) up to and including 30 days following coronary artery bypass graft (CABG) surgery compared with placebo.

DETAILED DESCRIPTION:
Coronary artery bypass grafting (CABG) effectively relieves angina, results in longer survival, and a better quality of life in specific subgroups of patients with obstructive coronary artery disease. Due to the high incidence of coronary artery disease worldwide, as well as the effectiveness of the surgical procedure, CABG surgery makes up one of the top ten most frequently performed procedures in North America and Europe. In the United States it is estimated that approximately 467,000 CABG procedures were performed in 2003.

Despite the benefits of CABG surgery, patients undergoing these procedures may also suffer serious adverse outcomes including operative mortality, myocardial infarction, unstable angina, ventricular failure, life-threatening arrhythmia, renal insufficiency, and stroke. Some of the proposed causes of cardiovascular morbidity and mortality after CABG include perioperative ischemia, inadequate myocardial protection and reperfusion injury. The impact of these serious complications is significant. Incidence rates of death and MI following CABG surgery range from 5% to 12% depending on risk status. Results from large clinical trials have recently demonstrated the importance of neurologic deficits as a problematic outcome of CABG. These deficits include memory impairment, psychomotor, visuospatial, attention and language abilities as measured by neuropsychological testing as well as sensorimotor abnormalities associated with stroke.

MC-1 is a naturally occurring metabolite of vitamin B6. Evidence from pre-clinical and clinical studies suggests that MC-1 protects the heart from ischemic damage and ischemia-reperfusion injury. This trial will assess the cardioprotective effects of MC-1 compared to placebo in patients undergoing high-risk CABG surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be scheduled to undergo CABG surgery (during routine scheduling times) and had planned to use cardiopulmonary bypass.
* Provide informed consent
* Age ≥ 18
* Male patients, or female patients not of childbearing potential or who have had a negative pregnancy test and are practicing adequate contraception
* Patients must be considered at high risk for subsequent myocardial complications defined as meeting 2 or more of the following:

  * Age ≥ 65
  * Current or recent smoker (within last 6 months)
  * History of diabetes mellitus requiring treatment other than diet
  * Evidence of left ventricular dysfunction or congestive heart failure assessed by:

    * Ejection fraction (EF) ≤ 45%
    * Left ventricular end diastolic pressure (LVEDP) or pulmonary wedge pressure (PWP) ≥ 20 mm Hg
    * Pulmonary edema by chest X-ray
    * Cardiothoracic ratio > 50% on chest X-ray
  * History of a previous non-disabling stroke, transient ischemic attack, or carotid endarterectomy
  * Urgent CABG intervention defined as the need to stay in the hospital (although patient may be operated on within a normal scheduling routine)
  * History of a myocardial infarction that occurred more than 48 hours but less than 6 weeks prior to CABG surgery
  * Prior peripheral artery surgery or angioplasty
  * Moderate renal dysfunction defined as creatinine clearance ≥ 30 ml/min, but < 60 ml/min
  * Presence of at least one asymptomatic carotid artery stenosis (≥ 50%) either in one or two carotid arteries

Exclusion Criteria:

* Planned associated valve surgery or concurrent carotid endarterectomy
* Planned aortic dissection repair or aortic root reconstruction
* Screening visit occurring less than 4 hours before scheduled CABG surgery
* Mini-Mental State Examination (MMSE) score less than 24 at the screening visit
* Current cardiogenic shock, acute left ventricular rupture, ventricular septal rupture, or papillary muscle rupture
* Uncontrolled diabetes defined as fasting serum blood glucose value equal to or greater than 24 mmol/L (432 mg/dl) at the time of screening (if fasting serum blood glucose not obtained at screening, values obtained within 30 days prior to screening visit may be used)
* Myocardial infarction occurring < 48 hours prior to planned CABG surgery
* Severe renal dysfunction defined as an estimated creatinine clearance value of < 30 ml/min or nephrotic syndrome at screening (or measured creatinine clearance value obtained within 30 days prior to screening visit)
* History of liver cirrhosis, chronic active hepatitis (known positive serum test within 6 months of enrolment), or severe liver dysfunction; or liver transaminase ≥ 3 times upper limit of normal (ULN) at screening (or obtained within 30 days prior to screening visit).
* History of malignancy during last 5 years except for basal cell carcinoma
* Planned surgery for atrial fibrillation
* Planned associated transmyocardial revascularization
* Planned associated ventricular remodeling
* Pregnancy or potential for pregnancy
* Any medical or psychiatric condition which, in the opinion of the investigator, makes the patient an unsuitable candidate for the study
* Significant, ongoing alcohol or drug abuse
* Participation in any other investigational drug or device study within 30 days of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2006-11; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
combined incidence of cardiovascular death or nonfatal myocardial infarction on days up to and including post-operative day (POD) 30

SECONDARY OUTCOMES:
length of hospital stay for index hospitalization
length of stay in intensive care unit (ICU) or coronary care unit (CCU) for index hospitalization
incidence of cardiovascular death up to and including POD 90

CONTACTS AND LOCATIONS:
Overall Officials: Michel Carrier, MD, Principal Investigator — Montreal Heart Institute; Robert A Harrington, MD, Principal Investigator — Duke Clinical Research Institute
Locations (2):
- Duke Clinical Research Institute, Durham, North Carolina, United States
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Background] Kandzari DE, Labinaz M, Cantor WJ, Madan M, Gallup DS, Hasselblad V, Joseph D, Allen A, Green C, Hidinger KG, Krucoff MW, Christenson RH, Harrington RA, Tcheng JE. Reduction of myocardial ischemic injury following coronary intervention (the MC-1 to Eliminate Necrosis and Damage trial). Am J Cardiol. 2003 Sep 15;92(6):660-4. doi: 10.1016/s0002-9149(03)00818-x. PMID 12972102
- [Derived] MEND-CABG II Investigators; Alexander JH, Emery RW Jr, Carrier M, Ellis SJ, Mehta RH, Hasselblad V, Menasche P, Khalil A, Cote R, Bennett-Guerrero E, Mack MJ, Schuler G, Harrington RA, Tardif JC. Efficacy and safety of pyridoxal 5'-phosphate (MC-1) in high-risk patients undergoing coronary artery bypass graft surgery: the MEND-CABG II randomized clinical trial. JAMA. 2008 Apr 16;299(15):1777-87. doi: 10.1001/jama.299.15.joc80027. Epub 2008 Apr 1. PMID 18381567
- [Derived] Mehta RH, Alexander JH, Emery R, Ellis SJ, Hasselblad V, Khalil A, Carrier M, Harrington RA, Tardif JC; MEND-CABG II Investigators. A randomized, double-blind, placebo-controlled, multicenter study to evaluate the cardioprotective effects of MC-1 in patients undergoing high-risk coronary artery bypass graft surgery: MC-1 to Eliminate Necrosis and Damage in Coronary Artery Bypass Graft Surgery Trial (MEND-CABG) II--study design and rationale. Am Heart J. 2008 Apr;155(4):600-8. doi: 10.1016/j.ahj.2008.01.002. Epub 2008 Feb 21. PMID 18371465